CLINICAL TRIAL: NCT04422210
Title: A Phase Ib Dose-Escalation and Dose-Expansion Study Evaluating The Safety, Tolerability, Pharmacokinetics, And Efficacy Of Venetoclax In Combination With Atezolizumab, Carboplatin, And Etoposide In Patients With Untreated Extensive-Stage Small Cell Lung Cancer.
Brief Title: A Study Evaluating The Safety, Tolerability, Pharmacokinetics, And Efficacy Of Venetoclax In Combination With Atezolizumab, Carboplatin, And Etoposide In Participants With Untreated Extensive-Stage Small Cell Lung Cancer (ES-SCLC).
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Decision to discontinue the study based on broader development and strategic prioritisation. The Sponsor concludes there is no benefit-risk impact on the GO41864 study.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO41864; 2019-004487-22 (EudraCT Number)
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Results first posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — venetoclax; atezolizumab; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Dose Escalation (Arm A1) (Maintenance only) (Experimental): Cohort A1: Participants with ES-SCLC who completed 4-6 cycles of carboplatin and etoposide first-line induction chemotherapy, with or without atezolizumab, were administered continuous maintenance therapy with Venetoclax (400mg) once daily (QD) from Day 1 to 21 and Atezolizumab (1200mg) every 3 weeks (Q3W) on Day 1.
  Interventions: Drug: Venetoclax; Drug: Atezolizumab
- Dose Escalation (Arm A2) (Maintenance only) (Experimental): Cohort A2: Participants with ES-SCLC who completed 4-6 cycles of carboplatin and etoposide first-line induction chemotherapy, with or without atezolizumab, were to be administered continuous maintenance therapy with Venetoclax (800mg) once daily (QD) from Day 1 to 21 and Atezolizumab (1200mg) every 3 weeks (Q3W) on Day 1.
  Interventions: Drug: Venetoclax; Drug: Atezolizumab
- Dose Escalation (Arm A3) (Maintenance only) (Experimental): Cohort A3: Participants with ES-SCLC who completed 4-6 cycles of carboplatin and etoposide first-line induction chemotherapy, with or without atezolizumab, were to be administered continuous maintenance therapy with Venetoclax (200mg) once daily (QD) from Day 1 to 21 and Atezolizumab (1200mg) every 3 weeks (Q3W) on Day 1. This cohort maybe explored if Dose-Limiting Toxicities (DLTs) are experienced and adverse events are thought to be potentially mitigated with a lower dose of venetoclax.
  Interventions: Drug: Venetoclax; Drug: Atezolizumab
- Dose Escalation (Arm B1) (Induction + Maintenance) (Experimental): Cohort B1: Participants with ES-SCLC were to be administered non-continuous induction therapy with Venetoclax (200mg) once daily (QD) from Day 1 to 7, Atezolizumab (1200mg) every 3 weeks (Q3W) on Day 1, Carboplatin (5mg/mL/min) on Day 1 and Etoposide (100mg/m^2) on Days 1-3. Participants who tolerated study treatment without excessive toxicity, and had not undergone disease progression were to be then proceeded to maintenance treatment with venetoclax plus atezolizumab. The venetoclax dose for the maintenance setting in Arm B will be the dose that has been cleared in the maintenance only arm (Arm A) of the study (maintenance RP2D, RP2D-M).
  Interventions: Drug: Venetoclax; Drug: Atezolizumab; Drug: Carboplatin; Drug: Etoposide
- Dose Escalation (Arm B2) (Induction + Maintenance) (Experimental): Cohort B2: Participants with ES-SCLC were to be administered non-continuous induction therapy with Venetoclax (400mg) once daily (QD) from Day 1 to 7, Atezolizumab (1200mg) every 3 weeks (Q3W) on Day 1, Carboplatin (5mg/mL/min) on Day 1 and Etoposide (100mg/m^2) on Days 1-3. Participants who tolerated study treatment without excessive toxicity, and had not undergone disease progression were to be then proceeded to maintenance treatment with venetoclax plus atezolizumab. The venetoclax dose for the maintenance setting in Arm B will be the dose that has been cleared in the maintenance only arm (Arm A) of the study (maintenance RP2D, RP2D-M).
  Interventions: Drug: Venetoclax; Drug: Atezolizumab; Drug: Carboplatin; Drug: Etoposide
- Dose Escalation (Arm B3) (Induction + Maintenance) (Experimental): Cohort B3: Participants with ES-SCLC were to be administered non-continuous induction therapy with Venetoclax (800mg) once daily (QD) from Day 1 to 7, Atezolizumab (1200mg) every 3 weeks (Q3W) on Day 1, Carboplatin (5mg/mL/min) on Day 1 and Etoposide (100mg/m^2) on Days 1-3. Participants who tolerated study treatment without excessive toxicity, and had not undergone disease progression were to be then proceeded to maintenance treatment with venetoclax plus atezolizumab. The venetoclax dose for the maintenance setting in Arm B will be the dose that has been cleared in the maintenance only arm (Arm A) of the study (maintenance RP2D, RP2D-M).
  Interventions: Drug: Venetoclax; Drug: Atezolizumab; Drug: Carboplatin; Drug: Etoposide
- Dose Escalation (Arm B4) (Induction + Maintenance) (Experimental): Cohort B4: Participants with ES-SCLC were to be administered non-continuous induction therapy with Venetoclax (800mg) once daily (QD) from Day 1 to 14, Atezolizumab (1200mg) every 3 weeks (Q3W) on Day 1, Carboplatin (5mg/mL/min) on Day 1 and Etoposide (100mg/m^2) on Days 1-3. Participants who tolerated study treatment without excessive toxicity, and had not undergone disease progression were to be then proceeded to maintenance treatment with venetoclax plus atezolizumab. The venetoclax dose for the maintenance setting in Arm B will be the dose that has been cleared in the maintenance only arm (Arm A) of the study (maintenance RP2D, RP2D-M).
  Interventions: Drug: Venetoclax; Drug: Atezolizumab; Drug: Carboplatin; Drug: Etoposide
- Dose Expansion (Experimental): If the Recommended Phase II Dose (RP2D) for Venetoclax during induction is established, then the dose-expansion cohort would continue to test venetoclax in both induction and maintenance. Participants would be administered non-continuous induction therapy with Venetoclax (RP2D-I/induction RP2D), Atezolizumab (1200mg) every 3 weeks (Q3W) on Day 1, Carboplatin (5mg/mL/min) on Day 1 and Etoposide (100mg/m^2) on Days 1-3 followed by continuous maintenance therapy with Venetoclax (RP2D-M) and Atezolizumab (1200mg) every 3 weeks (Q3W) on Day 1. If significant toxicity and DLTs in induction precluded identification of an RP2D for venetoclax in induction treatment, then the safety and efficacy of venetoclax would only be investigated in dose-expansion in the maintenance setting. Participants would be administered continuous maintenance therapy with Venetoclax (RP2D-M) and Atezolizumab (1200mg) every 3 weeks (Q3W) on Day 1.
  Interventions: Drug: Venetoclax; Drug: Atezolizumab; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Venetoclax — Venetoclax will be administered orally at escalating doses from 200mg to 800mg as 100mg tablets as per the dosing schedules described above.
Drug: Atezolizumab — Atezolizumab will be administered via intravenous (IV) infusion at a fixed dose of 1200mg as per the dosing schedules described above.
Drug: Carboplatin — Carboplatin will be administered via IV infusion at a dose of 5mg/mL/min as per the dosing schedules described above.
  Arms: Dose Escalation (Arm B1) (Induction + Maintenance); Dose Escalation (Arm B2) (Induction + Maintenance); Dose Escalation (Arm B3) (Induction + Maintenance); Dose Escalation (Arm B4) (Induction + Maintenance); Dose Expansion
Drug: Etoposide — Etoposide will be administered via IV infusion at a dose of 100mg/m^2 as per the dosing schedules described above.
  Arms: Dose Escalation (Arm B1) (Induction + Maintenance); Dose Escalation (Arm B2) (Induction + Maintenance); Dose Escalation (Arm B3) (Induction + Maintenance); Dose Escalation (Arm B4) (Induction + Maintenance); Dose Expansion

SUMMARY:
A study consisting of a dose-escalation phase and a dose-expansion phase to evaluate the safety, tolerability, pharmacokinetics, and efficacy of venetoclax in combination with atezolizumab, carboplatin, and etoposide.

ELIGIBILITY:
Inclusion Criteria:

Dose Escalation, Maintenance Arm A:

* Participants with ES-SCLC who have completed 4-6 cycles of carboplatin and etoposide induction chemotherapy, with or without atezolizumab, as their first-line therapy for extensive-stage disease and have responded (CR or PR) or have Stable Disease (SD) are eligible for the maintenance arm of the study.
* All side effects attributed to prior anti-cancer therapy must have resolved to Grade 1 or baseline.
* A maximum of 8 weeks (56 days) is allowed between last chemotherapy dose (Cycle 4, Day 3) given in induction and the start of maintenance therapy.

Dose Escalation, Induction Arm B:

* Participants with no prior systemic treatment for ES-SCLC are eligible for this study.
* ANC >= 1,500 cells/µL without granulocyte colony-stimulating factor support.

Dose Expansion, Maintenance-Only:

* Participants with ES-SCLC who have completed 4 cycles of carboplatin and etoposide induction chemotherapy and at least 3 cycles of atezolizumab as their first-line therapy for extensive-stage disease and have responded (CR or PR) or have SD are eligible for the maintenance arm of the study.

Dose Escalation (Arms A and B) and Dose Expansion:

* Ability to comply with the study protocol, in the investigator's judgement.
* ECOG performance status of 0 or 1.
* Participants must be able to swallow pills.
* Histologically or cytologically confirmed diagnosis of ES-SCLC per the Veterans Administration Lung Study Group (VALG) staging system.
* Participants who received prior chemoradiotherapy for limited-stage SCLC must have been treated with curative intent and experienced a treatment-free interval of at least 6 months since last chemotherapy, radiotherapy or chemoradiotherapy cycle prior to diagnosis of ES-SCLC.
* Participants with a history of treated CNS metastases that are currently asymptomatic.
* Measurable disease, as defined by RECIST v1.1. Baseline measurements and evaluation of all sites of disease must be obtained =<4 weeks prior to enrollment.
* Eligible to receive a carboplatin-based chemotherapy regimen.
* Adequate hematologic and end-organ function.
* Participants must submit a pre-treatment tumor tissue sample.
* Participants must submit a blood sample for exploratory biomarker research before treatment, on-study, and following progression of disease.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse), use non-hormonal contraceptive methods and refrain from donating eggs.
* Women who are not postmenopausal (>=12 months of non-therapy-induced amenorrhea) or surgically sterile must have a negative serum pregnancy test result within 14 days prior to initiation of study drug.
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom and agreement to refrain from donating sperm.

Exclusion Criteria:

* Use of non-protocol-specified anti-cancer therapies or other combination partners with carboplatin/etoposide during induction.
* Symptomatic or actively progressing CNS metastases.
* Pregnant or breastfeeding, or intending to become pregnant during the study.
* Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for >= 1 week prior to enrollment.
* Leptomeningeal disease.
* Uncontrolled pleural effusion, pericardial effusion or ascites requiring recurrent drainage procedures (once a month or more frequently).
* Uncontrolled or symptomatic hypercalcemia.
* History of malignancy other than SCLC within 5 years prior to enrollment.
* History of autoimmune disease.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
* Positive HIV infection.
* Active Hepatitis B and C infection (HBV/HCV).
* Active Tuberculosis infection.
* Known infection with human T-cell leukemia virus 1.
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment, or any major episode of infection requiring treatment with IV antibiotics or hospitalization.
* Significant cardiovascular disease.
* Major surgical procedure within 28 days prior to enrollment or anticipation of need for major surgical procedure during the course of the study.
* Prior allogenic bone marrow transplantation or solid organ transplant.
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the participant at high risk for treatment complications.
* Illnesses or conditions that interfere with their capacity to understand, follow, and/or comply with study procedures.
* Treatment with investigational therapy with therapeutic intent within 28 days prior to enrollment.
* Administration of a live, attenuated vaccine within 4 weeks before enrollment or anticipation that such a live attenuated vaccine will be required during the study.
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, anti-PD-1, and anti-PD-L1 therapeutic antibodies.
* Treatment with systemic immunosuppressive medications within 1 week prior to enrollment.
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
* Known hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation.
* History of allergic reactions to carboplatin or etoposide or to any of its excipients (etoposide).
* Known hypersensitivity to venetoclax or to any of its excipients.
* Administration of Steroid therapy for anti-neoplastic intent, strong or moderate CYP3A inhibitors or strong or moderate CYP3A inducers within 7 days prior to the first dose of study drug.
* Consumption of grapefruit, grapefruit products, Seville oranges (including marmalade-containing Seville oranges), or starfruit (carambola) within 3 days prior to the first dose of study drug.
* Malabsorption syndrome or other condition that would interfere with enteral absorption.
* Illicit drug or alcohol abuse within 12 months prior to screening, in the investigator's judgement.
* Inability or unwillingness to swallow a large number of tablets.
* History of inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis) or active bowel inflammation (e.g., diverticulitis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- Emory University, Atlanta, Georgia, United States
- Rigshospitalet; Onkologisk Klinik, København Ø, Denmark
- Severance Hospital, Yonsei University Health System, Seoul, South Korea
- Spain (2):
  - ICO I Hospitalet Hospital Duran i Reynals Instituto Catalan de Oncologia de Hospitalet ICO, L'Hospitalet de Llobregat, Barcelona
  - START Madrid. Centro Integral Oncologico Clara Campal; CIOCC, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated by the Sponsor. Only 2 participants were enrolled in this study. Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Period: Overall Study
Arm/Group | Dose Escalation (Arm A1) (Maintenance Only) | Dose Escalation (Arm A2) (Maintenance Only) | Dose Escalation (Arm A3) (Maintenance Only) | Dose Escalation (Arm B1) (Induction + Maintenance) | Dose Escalation (Arm B2) (Induction + Maintenance) | Dose Escalation (Arm B3) (Induction + Maintenance) | Dose Escalation (Arm B4) (Induction + Maintenance) | Dose Expansion
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated by the Sponsor. Only 2 participants were enrolled in this study. Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation (Arm A1) (Maintenance Only) | Dose Escalation (Arm A2) (Maintenance Only) | Dose Escalation (Arm A3) (Maintenance Only) | Dose Escalation (Arm B1) (Induction + Maintenance) | Dose Escalation (Arm B2) (Induction + Maintenance) | Dose Escalation (Arm B3) (Induction + Maintenance) | Dose Escalation (Arm B4) (Induction + Maintenance) | Dose Expansion | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [unit: years]
Sex: Female, Male [unit: Participants]
Race/Ethnicity, Customized [unit: Participants]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: The study was terminated by the Sponsor. Only 2 participants were enrolled in this study. Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: Baseline up until 30 days after the last dose of study drug or until initiation of new systemic anti-cancer therapy, whichever occurs first (up to a maximum of 6.5 weeks).
Population: as for baseline characteristics
Arm/Group | Dose Escalation (Arm A1) (Maintenance Only) | Dose Escalation (Arm A2) (Maintenance Only) | Dose Escalation (Arm A3) (Maintenance Only) | Dose Escalation (Arm B1) (Induction + Maintenance) | Dose Escalation (Arm B2) (Induction + Maintenance) | Dose Escalation (Arm B3) (Induction + Maintenance) | Dose Escalation (Arm B4) (Induction + Maintenance) | Dose Expansion
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Overall Response Rate (ORR)
Description: as for outcome 1
Time Frame: Up to 24 months
Population: as for baseline characteristics
Arm/Group | Dose Expansion
Number analyzed (Participants) | 0

3. Secondary Outcome: Duration of Response (DOR)
Description: as for outcome 1
Time Frame: Up to 24 months
Population: as for baseline characteristics
Arm/Group | Dose Expansion
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression Free Survival (PFS)
Description: as for outcome 1
Time Frame: Up to 24 months
Population: as for baseline characteristics
Arm/Group | Dose Expansion
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival (OS) After Enrolment
Description: as for outcome 1
Time Frame: Up to 49 months
Population: as for baseline characteristics
Arm/Group | Dose Expansion
Number analyzed (Participants) | 0

6. Secondary Outcome: Progression Free Survival (PFS) Rate at 6 Months
Description: as for outcome 1
Time Frame: Up to 18 months
Population: as for baseline characteristics
Arm/Group | Dose Expansion
Number analyzed (Participants) | 0

7. Secondary Outcome: Overall Survival (OS) Rate at 1 Year
Description: as for outcome 1
Time Frame: Up to 18 months
Population: as for baseline characteristics
Arm/Group | Dose Expansion
Number analyzed (Participants) | 0

8. Secondary Outcome: Plasma Concentrations (ng/mL) of Venetoclax at Specified Timepoints
Description: as for outcome 1
Time Frame: Up to 24 months
Population: as for baseline characteristics
Arm/Group | Dose Escalation (Arm A1) (Maintenance Only) | Dose Escalation (Arm A2) (Maintenance Only) | Dose Escalation (Arm A3) (Maintenance Only) | Dose Escalation (Arm B1) (Induction + Maintenance) | Dose Escalation (Arm B2) (Induction + Maintenance) | Dose Escalation (Arm B3) (Induction + Maintenance) | Dose Escalation (Arm B4) (Induction + Maintenance)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Serum Concentrations (ng/mL) of Atezolizumab at Specified Timepoints
Description: as for outcome 1
Time Frame: Up to 24 months
Population: as for baseline characteristics
Arm/Group | Dose Escalation (Arm A1) (Maintenance Only) | Dose Escalation (Arm A2) (Maintenance Only) | Dose Escalation (Arm A3) (Maintenance Only) | Dose Escalation (Arm B1) (Induction + Maintenance) | Dose Escalation (Arm B2) (Induction + Maintenance) | Dose Escalation (Arm B3) (Induction + Maintenance) | Dose Escalation (Arm B4) (Induction + Maintenance)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Plasma Concentrations (ng/mL) of Carboplatin at Specified Timepoints
Description: as for outcome 1
Time Frame: Up to 24 months
Population: as for baseline characteristics
Arm/Group | Dose Expansion
Number analyzed (Participants) | 0

11. Secondary Outcome: Plasma Concentrations (ng/mL) of Etoposide at Specified Timepoints
Description: as for outcome 1
Time Frame: Up to 24 months
Population: as for baseline characteristics
Arm/Group | Dose Expansion
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The study was terminated by the Sponsor. Only 2 participants were enrolled in this study. Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Description: The study was terminated by the Sponsor. Only 2 participants were enrolled in this study. Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Arm/Group | Dose Escalation (Arm A1) (Maintenance Only) | Dose Escalation (Arm A2) (Maintenance Only) | Dose Escalation (Arm A3) (Maintenance Only) | Dose Escalation (Arm B1) (Induction + Maintenance) | Dose Escalation (Arm B2) (Induction + Maintenance) | Dose Escalation (Arm B3) (Induction + Maintenance) | Dose Escalation (Arm B4) (Induction + Maintenance) | Dose Expansion
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated by the Sponsor. Only 2 participants were enrolled in this study. Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/10/NCT04422210/Prot_SAP_000.pdf